CLINICAL TRIAL: NCT05413733
Title: Feasibility and Effectiveness of Web-based Neuropsychological Rehabilitation After Acquired Brain Injury
Brief Title: Neuropsychological Rehabilitation Over the Internet
Acronym: IRENE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Eeva-Liisa Kallio, Neuropsychologist, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TYH2022304
Record Dates: First submitted 2022-05-28; First posted 2022-06-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Acute Ischemic; Brain Hemorrhage; Encephalitis; Hypoxia-Ischemia, Brain; Traumatic Brain Injury
Keywords: web-based intervention; neuropsychological rehabilitation; psychoeducation; acquired brain injury
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages; Encephalitis; Hypoxia-Ischemia, Brain; Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Intervention Model Description: A parallel-group randomized controlled trial
Who Masked: Care Provider
Masking Description: Digital care pathway is part of the daily neurological treatment at HUS. Care providers will be clinical neuropsychologists who do not know if their patient is involved in the study or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital care pathway (Experimental): Intervention group goes through a web-based neuropsychological intervention program. The program includes eight structured sessions regarding general neuropsychological symptoms after ABI - problems with fatigue, attention, executive functions and memory. A new session opens after the previous one is completed, and after a minimum of 3 days between the sessions. The intervention takes approximately 2 months depending on the progression pace of a patient. The eight sessions consist of psychoeducation, self-assessments, cognitive strategy training and feedback (automatic or given by a monitoring neuropsychologist). A neuropsychologist from HUS monitors patients' progression and provides personal feedback when needed. Participants can also be in contact with a monitoring neuropsychologist via message feature of the program.
  Interventions: Behavioral: Digital care pathway
- Care as usual (Active Comparator): Control group attends the standard care of patients with ABI in HUS including all necessary outpatient rehabilitation visits. When available, neuropsychological rehabilitation typically takes 1-2 months among the study target group.
  Interventions: Behavioral: Care as usual

INTERVENTIONS:
Behavioral: Digital care pathway — Sessions of the digital neuropsychological program:
  1. Subjective functional ability and goals
  2. Fatigue after ABI
  3. Attention and concentration
  4. Memory
  5. Memory strategies
  6. Working memory and executive functions
  7. Emotional reactions
  8. Summary and future goals
  Other Names: iRENE Digital pathway
  Arms: Digital care pathway
Behavioral: Care as usual — The standard care of patients with ABI including all necessary outpatient rehabilitation visits. Neuropsychological visits may include a short period of psychoeducation with a clinical neuropsychologist.
  Arms: Care as usual

SUMMARY:
Helsinki University Hospital (HUS) has decided on a strategy to provide digital health care services for several medical specialties - a project called the Health Village (HealthVillage.fi). Within Health Village a specific digital My Path program, iRENE Digital Pathway, has been developed for web-based neuropsychological rehabilitation. iRENE Digital Pathway is a structured program for adults with an acquired brain injury (ABI), which utilizes psychoeducative information and self-evaluation questionnaires for attentional, memory and executive disorders with a feedback, and provides training for internal and external memory and other cognitive strategies. The current study will explore if web-based neuropsychological rehabilitation is a feasible and effective method for carrying out rehabilitation for adults with ABI.

DETAILED DESCRIPTION:
The IRENE study will explore the application, feasibility and effectiveness of web-based neuropsychological rehabilitation for working-aged patients with ABI during the first year of recovery. This study will adopt a 2-arm randomized controlled design with treatment-as-usual control.

The investigators will determine the feasibility and effectiveness of a web-based rehabilitation program for patients with ABI on their subjective memory difficulties, management of cognitive symptoms, self-efficacy, fatigue, mood, anxiety, quality of life and subjective working ability. The study will examine, if the method is accessible as well as if neurological patients are able and willing to use web-based rehabilitation. The potential health-economic benefits of the new rehabilitation program will be assessed with the duration of patients' sick leave after ABI and through the net benefit of neuropsychological rehabilitation resources.

A pilot randomized trial with 60 participants will be conducted to address the rate of recruitment of the participants, patient acceptability and adherence to study protocol, retention rates and feedback of the iRENE program as well as initial data on effectiveness of this new program. This pilot trial will use an unequal randomization 2:1 to maximize experiences in delivering the digital intervention to patients after ABI. The intervention group will participate in the iRENE Digital Pathway, a web-based rehabilitation program, that takes 2-3 months to complete. The control group attends treatment as usual, which includes necessary outpatient rehabilitation.

Outcome measures at baseline, post-intervention and 3-month follow-up after completing the intervention are gathered as self-assessments.

The participants are adult patients from neurological acute wards and outpatient clinics from HUS, Finland. Patients with ABI typically get referral to neuropsychological examination at the acute or the sub-acute phase of recovery. The examining clinical neuropsychologist offers a patient the possibility to get involved in the research. A neuropsychologist from the research group interviews voluntary patients at hospital or via telephone to confirm patient's interest and fulfillment of inclusion criteria.

Intervention group will go through a systematic web-based neuropsychological intervention program. Participants carry out the web-based intervention independently with their own digital appliance (computer, tablet or mobile phone) time and place of one's choice.

Control group attends the standard care of patients with ABI including all necessary outpatient rehabilitation visits. A possibility to attend to the iRENE Digital Pathway will be offered to control group participants after they have performed the 5-month assessment of the study.

ELIGIBILITY:
Inclusion Criteria:

* Acute neurological incident affecting cognition (stroke, encephalitis, traumatic brain injury, anoxia)
* Less than 6 months from occurrence of an acute neurological incident
* Mild to moderate cognitive deficits on a clinical neuropsychological assessment during inpatient or outpatient care after ABI
* Subjective cognitive symptoms following ABI
* Proficient in Finnish
* Must be able to use digital appliances

Exclusion Criteria:

* Not an acute neurological incident
* More than 6 months from an acute neurological incident
* Severe cognitive deficits on a clinical neuropsychological assessment during inpatient or outpatient care after ABI
* Not fluent in Finnish
* Not able to use digital appliances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Baseline Perceived Subjective Cognitive symptoms at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the Everyday Memory Questionnaire - Revised; The minimum total score is 0 and the maximum score is 52; The higher total score represents more severe subjective cognitive symptoms

SECONDARY OUTCOMES:
Change of Baseline Perceived Use of Memory Aids at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the Adaptation to Memory Difficulties Outcome Questionnaire; The questionnaire includes subscales assessing memory knowledge and emotional adjustment (15 questions), use of external memory aids (5 questions) and use of internal memory aids (5 questions); Each item will be scored on a 4-point scale 1-4; Each of the three parts of the questionnaire will be analyzed separately; A higher score would signify better adaptation.
Change of Baseline Perceived Self-Efficacy at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the New General Self-Efficacy Scale; The New General Self-Efficacy Scale is an 8-item measure that assesses how much people believe they can achieve their goals, despite difficulties; The minimum total score is 1 and the maximum score is 5; The higher total score represents higher self-efficacy
Change of Baseline Perceived Anxiety at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the Patient-Reported Outcomes Measurement Information System (PROMIS): anxiety; The minimum total raw score is 8 and the maximum score is 40; The higher total score represents higher anxiety
Change of Baseline Perceived Depression at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the Patient-Reported Outcomes Measurement Information System (PROMIS): depression; The minimum total raw score is 8 and the maximum score is 40; The higher total score represents higher depression
Change of Baseline Perceived Quality of life at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the Euro-Qol (EQ-5D) Questionnaire; The minimum total raw score is 0 and the maximum score is 100; The higher score represents higher quality of life in terms of self-perceived health
Change of Baseline Perceived Fatigue at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the Fatigue Assessment Scale; The minimum total raw score is 10 and the maximum score is 50; The higher total score represents more severe fatigue

OTHER OUTCOMES:
Change of Baseline Perceived Working ability at 2 months and 5 months | Baseline, Month 2, and Month 5
  Administration of the Work Ability Index; The minimum total score is 0 and the maximum score is 24; The higher total score represents better self-perceived working ability
Length of sick leave of a patient | Month 5
  Length of sick leave in days after acquired brain injury
Intervention feedback questionnaire | Month 2
  Feedback of the neuropsychological rehabilitation period offered during the study; Participants give their evaluation in a 5-point likert scale; The higher total score represents more positive evaluation;
  % of patients with positive and negative evaluation will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Marja Hietanen, PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- HUS Neurocenter, Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Short introduction to My Path in Health Village — https://www.terveyskyla.fi/en/mypath